CLINICAL TRIAL: NCT03133949
Title: Aortitis and Retroperitoneal Fibrosis: Evaluation of Diagnostic Criteria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PHRCIR09-DR-SCHMIDT
Record Dates: First submitted 2017-04-13; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Aortitis; Retroperitoneal Fibrosis
MeSH Terms: conditions — Retroperitoneal Fibrosis | interventions — Biological Products

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with idiopathic inflammatory aortitis
  Interventions: Other: Establish the clinical, biological and radiological characteristics of patients
- a group of witnesses
  Interventions: Other: Establish the clinical, biological and radiological characteristics of patients

INTERVENTIONS:
Other: Establish the clinical, biological and radiological characteristics of patients — Establish the clinical, biological and radiological characteristics of patients

SUMMARY:
Inflammatory aortitis probably represents a heterogeneous group, and the clinical experience accumulated over the last ten years, shared by the experts of the subject, is that the initial clinical, biological or radiological characteristics should make it possible to differentiate them and dismember the Nosological field.

This will be an essential first step before studying prognosis, risk factors, and therapeutic options.

The search for diagnostic criteria on a large series, similar to the study of classification of vascularites of the ACR in 1990, should make it possible to homogenize the diagnoses for the different teams working on the subject, and to begin work Collaborations, which alone can improve patient care in the future.

ELIGIBILITY:
Inclusion Criteria:

* Cases :

  * All cases of idiopathic aortitis and retroperitoneal fibrosis followed in participating centers over the past 15 years will be collected.
* Witnesses :

  * Group 1: non-idiopathic inflammatory aortitis: all cases of inflammatory aortitis (apart from idiopathic aortites and isolated retroperitoneal fibrosis) followed in the participating centers over the last 15 years will be collected.
  * Group 2: subjects with noninflammatory aortic disease, atheromatous type or annulo-ectasitic disease, matched by age and sex with cases. This group will be used to define the differential characteristics between idiopathic aortitis and noninflammatory aortic pathology.
  * Group 3: This group will include control subjects aimed at defining radiological normality criteria according to age and sex. As the images are machine-dependent, group 3 controls will be randomly selected from the radiology departments that have performed the scanner or MRI of the corresponding control.

Exclusion Criteria:

* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with idiopathic inflammatory aortitis or retroperitoneal fibrosis.
  Three focus groups will be constituted:
  Group 1: it will include all cases of non-idiopathic inflammatory aortitis followed in the participating centers over the last 15 years, Group 2: it will include patients with non-inflammatory aortic conditions (aneurysm, atheroma, annulo-ectasitic aortic disease).
  Group 3: it will include patients without aortic pathology matched by age and sex, having a thoracoabdominal scanner or MRI in the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2010-07-08 (Actual); Primary Completion 2020-07-08 (Estimated); Study Completion 2020-07-08 (Estimated)

PRIMARY OUTCOMES:
Analyze the management of patients with aortic and retroperitoneal fibrosis | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France